CLINICAL TRIAL: NCT01716104
Title: Multicentric Double-blind Placebo-controlled Randomized Parallel-group Clinical Trial of Safety and Efficacy of Afalaza in Patients With Symptoms of Benign Prostatic Hyperplasia and Risk of Progression
Brief Title: Clinical Trial of Safety and Efficacy of Afalaza in Patients With Symptoms of Benign Prostatic Hyperplasia and Risk of Progression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-AZ-001-I
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afalaza (2 tablets twice a day) (Experimental)
  Interventions: Drug: Afalaza
- Placebo (2 tablets twice a day) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afalaza — Safety and Efficacy
  Arms: Afalaza (2 tablets twice a day)
Drug: Placebo — Safety and Efficacy
  Arms: Placebo (2 tablets twice a day)

SUMMARY:
The purpose of this study is:

* To assess safety of Afalaza drug within 12 months in patients with symptoms of benign prostatic hyperplasia (BPH) and risk of progression.
* To assess efficacy of Afalaza drug within 12 months in patients with symptoms of benign prostatic hyperplasia and risk of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients 45 to 60 y.o. inclusive with a documented diagnosis of Benign prostatic hyperplasia.
2. Lower urinary tract symptoms (LUTS) having been experienced for 3 months and longer.
3. Total IPSS score (International Prostate Symptome Score) of 8 to 15.
4. Prostate volume of more than 30 cm3.
5. Maximal urinary flow rate of 10-15 mL/sec.
6. Micturition volume of 125-350 mL.
7. Residual volume of less than 100 mL.
8. Serum prostate-specific antigen (PSA) level of less than 4 ng/mL.
9. Use of and compliance with contraceptive methods during the trial and for 30 days upon completion of participation in the trial.
10. Presence of the patient's information sheet (informed consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Invasive therapies for BPH including a transurethral prostatic resection, thermotherapy, microwave therapy, transurethral needle ablation, stenting, etc.
2. Malignant oncological disease of the urogenital system as well as malignancies of any other localization during last 5 years.
3. Acute urinary retention (AUR) within 3 months before inclusion in the trial.
4. Neurogenic dysfunctions and bladder ears.
5. Urinary stone disease.
6. Urethral stricture, bladder neck sclerosis.
7. History of operative aids for pelvic organs.
8. Urogenital infections in the phase of active inflammation.
9. Systematic administration of agents exhibiting effects on bladder function and urine production.
10. Exacerbation or decompensation of chronic diseases affecting the possibility of patients to participate in the clinical trial, including severe concurrent cardiovascular conditions and disorders of the nervous system, renal and hepatic insufficiency.
11. History of administration of testosterone 5-alpha-reductase inhibitors (finasteride, dutasteride).
12. History of polyvalent allergy.
13. Allergy/intolerance to any component of drug agents used in the therapy.
14. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency.
15. Administration of drugs specified as "Prohibited concomitant therapy", within 3 months before enrollment.
16. Exacerbation or decompensation of chronic diseases affecting the possibility of patients to participate in the clinical trial.
17. Drug and alcohol consumption (over 2 alc. units daily), mental diseases. Legal incapacity or limited legal capacity.
18. Legal incapacitation or limited legal capacity.
19. Patients, who, in the investigator's opinion, will fail to observe the requirements during the trial or adhere to the studied drug administration procedure.
20. Participation in other clinical trials within 3 months before enrolment in this trial.
21. Presence of other factors, complicating the patient's participation in the trial (e.g., planned lengthy business and other trips).
22. A patient is a part of the center's research staff, taking a direct part in the trial, or an immediate family member of the investigator. Immediate family members are defined as spouses, parents, children or siblings, regardless of whether full blood or adopted.
23. The patient is employed with Scientific Production Firm Materia Medica Holding LLC, i.e. is the company's employee, part-time employee under contract, or appointed official in charge of the trial, or their immediate family.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (15):
  - The State Budget Health Care institution of Moscow the City "Hospital for veterans of wars No. 2 of the Administration of Health Care of Moscow City", Moscow
  - The State Budget Health Care institution of Moscow the City "Specialized clinical (neuro-psychiatric) hospital No. 8 n.a. Z.P. Solovyov - ''Clinic of neuroses" of the Administration of Health Care of Moscow City, Moscow
  - The Federal State Budget Educational institution of High Professional Training "Peoples' Friendship University of Russia", Department of Urology and Operative Nephrology, Moscow
  - The State Budget Educational institution of High Professional Training I.M. Sechenov First Moscow State Medical University of Ministry of Health Care and Social Development of the Russian Federation, Department of Urology, Moscow
  - The State Budgetary Educational Institution of Higher Professional Education " Moscow State University of Medicine and Dentistry of A. I. Evdokimov" Ministry of Health of the Russian Federation, Moscow
  - The Federal State Budget institution "Polyclinic № 3" of Affairs Management Department of the President of the Russian Federation, Moscow
  - Limited liability company "Family Policlinic No. 4", Moscow Region Koroljov
  - Municipal Treatment-and-Prophylactic Health Care institution Clinical Diagnostic Centre "Zdorovie", Rostov-on-Don
  - The Federal State Budgetary Institution " Saint-Petersburg Research Institute Phthisiopulmonology " Ministry of Health of the Russian Federation, Saint Petersburg
  - The Federal State institution "All-Russian center of emergency and radiation medicine n.a. A.M. Nikiforov" of the Ministry of the Russian Federation for Affairs of civil defence, emergencies and elimination of consequences of natural disasters, Saint Petersburg
  - The Federal State Budgetary Health Care Institution "Clinical Hospital №122 n. a. L. G. Sokolov of the Federal Biomedical Agency", Saint Petersburg
  - Limited liability company "Medical unit No. 157", Saint Petersburg
  - Saint-Petersburg State Budget Health Care institution "Pokrovsky city hospital", Saint Petersburg
  - Limited Liability Company "Hospital OrCli", Saint Petersburg
  - The State Budgetary Educational Institution of Higher Professional Education " Siberian state Medical University" Ministry of Health of the Russian Federation, Tomsk
- The State Institution "Institute of Urology of the Ukraine National Academy of Medical Sciences", Kyiv, Ukraine

REFERENCES:
- [Derived] Pushkar D, Vinarov A, Spivak L, Kolontarev K, Putilovskiy M, Andrianova E, Epstein O. Efficacy and safety of Afalaza in men with symptomatic benign prostatic hyperplasia at risk of progression: a multicenter, double-blind, placebo-controlled, randomized clinical trial. Cent European J Urol. 2018;71(4):427-435. doi: 10.5173/ceju.2018.1803. Epub 2018 Dec 27. PMID 30680237

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Selection procedures were carried out after participant enrollment to determine whether the patient could participate in the study in accordance with the inclusion criteria.
  Of the 260 patients enrolled, 11 did not meet inclusion criteria after screening procedures, they were not randomized.
Groups:
- Afalaza: Afalaza (2 tablets twice a day) One tablet contains: affinity purified antibodies to endothelial nitric oxide synthase - 0.006g*, affinity purified antibodies to prostate-specific antigen - 0.006g*.
  *applied onto isomalt crystals as a mixture of three active aqueous-alcoholic dilutions of the drug substance - diluted 100^12, 100^30, 100^50 times, respectively.
  Excipients: lactose monohydrate; microcrystalline cellulose; magnesium stearate.
- Placebo: Placebo (2 tablets twice a day)
Period: Overall Study
Arm/Group | Afalaza | Placebo
Started | 125 | 124
Completed | 119 | 117
Not Completed | 6 | 7
Not completed — Do not meet inclusion criteria | 6 | 7

BASELINE CHARACTERISTICS:
Population: Intention to treat set
Groups:
- Afalaza: Afalaza (2 tablets twice a day): Safety and Efficiency
- Placebo: Placebo (2 tablets twice a day): Safety and Efficiency
- Total: Total of all reporting groups
Arm/Group | Afalaza | Placebo | Total
Number analyzed (Participants) | 119 | 117 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (4.2) | 54.4 (4.4) | 54.4 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 119 | 117 | 236
Region of Enrollment [Number; unit: participants]
  Ukraine | 1 | 3 | 4
  Russia | 118 | 114 | 232

OUTCOME MEASURES:

1. Primary Outcome: Change in Total IPSS Scores (International Prostate Symptome Score) After 1, 3, 6 and 12 Months Compared to Baseline.
Description: The International Prostate Symptom Score (IPSS) is based on the answers to 7 questions concerning urinary symptoms plus one question concerning quality of life (QoL). Each of the seven symptoms includes the assignment of scores from 0 to 5. The total score can therefore range from 0 to 35 points (asymptomatic to very symptomatic). The patient's quality of life (QoL) was evaluated separately in this clinical study.
Time Frame: Baseline, 1, 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Afalaza: Afalaza (2 tablets twice a day): Safety and Efficacy
- Placebo: Placebo (2 tablets twice a day): Safety and Efficacy
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
Scores on a scale
  Month 1 | -1.3 (1.7) | -0.6 (1.3)
  Month 3 | -2.3 (2.1) | -1.5 (1.9)
  Month 6 | -3.0 (2.5) | -1.9 (2.5)
  Month 12 | -3.7 (3.0) | -2.9 (2.4)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0005, Mixed Models Analysis

2. Secondary Outcome: Change in Dynamics of Irritative Symptoms Evaluated by IPSS (International Prostate Symptome Score) After 1, 3, 6 and 12 Months Compared to Baseline
Description: The International Prostate Symptom Score (IPSS) is based on the answers to 7 questions concerning urinary symptoms plus one question concerning quality of life (QoL). Each of the seven symptoms includes the assignment of scores from 0 to 5. The total score can therefore range from 0 to 35 points (asymptomatic to very symptomatic). The patient's quality of life (QoL) was evaluated separately in this clinical study.
  The sum of IPSS questions 2, 4, and 7 related to irritative symptoms. The total score of irritative symptoms can therefore range from 0 to 15 points (asymptomatic to very symptomatic).
Time Frame: Baseline and 1, 3, 6, 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
Scores on a scale
  Month 1 | -0.5 (0.9) | -0.3 (1.1)
  Month 3 | -0.9 (1.2) | -0.6 (1.2)
  Month 6 | -1.3 (1.5) | -0.8 (1.4)
  Month 12 | -1.5 (1.6) | -1.3 (1.5)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.035, Mixed Models Analysis

3. Secondary Outcome: Change in Maximum Urinary Flow Rate After 1, 3, 6 and 12 Months Compared to Baseline
Time Frame: Baseline and 1, 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
ml/s
  Month 1 | 1.3 (3.2) | 0.2 (2.6)
  Month 3 | 1.5 (3.2) | 0.7 (3.3)
  Month 6 | 1.7 (3.2) | 0.5 (2.7)
  Month 12 | 2.5 (4.3) | 1.4 (3.3)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0008, Mixed Models Analysis

4. Secondary Outcome: Change in Average Urinary Flow Rate After 1, 3, 6 and 12 Months Compared to Baseline
Time Frame: Baseline and 1, 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
ml/s
  Month 1 | 0.9 (2.0) | 0.2 (1.9)
  Month 3 | 1.3 (2.1) | 0.7 (2.5)
  Month 6 | 1.4 (2.0) | 0.5 (2.2)
  Month 12 | 1.4 (2.2) | 0.6 (2.5)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0011, Mixed Models Analysis

5. Secondary Outcome: Percent Change in Mean Values of Prostate Gland Volume at 3, 6 and 12 Months Compared to Baseline
Description: Change in the volume of the prostate gland as a percentage of the baseline according to transrectal ultrasound
Time Frame: Baseline and 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: percentage of prostate gland volume
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
percentage of prostate gland volume
  Month 3 | -6.6 (13.1) | -2.9 (12.5)
  Month 6 | -10.0 (13.4) | -4.9 (14.1)
  Month 12 | -11.8 (16.0) | -6.5 (14.7)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0054, Mixed Models Analysis

6. Secondary Outcome: Change in Mean Values of Micturition Volume at 3, 6 and 12 Months Compared to Baseline
Time Frame: Baseline and 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
ml
  Month 3 | 14.6 (105.0) | 1.4 (76.8)
  Month 6 | 27.5 (96.6) | 5.0 (88.4)
  Month 12 | 17.9 (106.0) | 0.4 (71.2)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0437, Mixed Models Analysis

7. Secondary Outcome: Change in the Mean Values of Residual Urine Volume at 3, 6 and 12 Months Compared to Baseline
Description: according to transabdominal ultrasound
Time Frame: Baseline and 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
ml
  Month 3 | -6.5 (26.5) | -0.9 (21.6)
  Month 6 | -8.8 (28.1) | -4.3 (20.9)
  Month 12 | -8.0 (30.1) | -3.5 (26.9)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0862, Mixed Models Analysis

8. Secondary Outcome: Change in Quality of Life (QoL Index of IPSS) at 3, 6 and 12 Months Compared to Baseline
Description: Quality of life (QoL) Due to Urinary Symptoms is an eight point of the IPSS scale referred to the patient's quality of life. The answers to this question range from "delighted" to "terrible" or 0 to 5.
Time Frame: Baseline and 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
Scores on a scale
  Month 3 | -0.4 (0.8) | -0.4 (0.7)
  Month 6 | -0.7 (0.8) | -0.5 (1.0)
  Month 12 | -1.0 (1.0) | -0.6 (1.2)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0621, Mixed Models Analysis

9. Secondary Outcome: Change in Total Value of Risk Factors for Progression (Total Score of IPSS, Prostate Volume, PSA Level, Maximum Urinary Flow Rate, Residual Urine Volume) Compared to Baseline
Description: To assess the risk of BPH progression, the following were used: 1) moderate to severe BPH symptoms (ie, IPSS total score> 7); 2) an increase in the volume of the prostate gland (> 30 cm^2); 3) increased PSA level in the blood (≥ 1.4 ng / ml); 4) a decrease in Qmax (<12 ml / s) and 5) a large volume of residual urine (> 200 ml).
  The total value of risk factors for progression is assessed as the sum of the risk factors that the patient had at the time of inclusion in the study (presence of risk factors = 1 point, absence = 0 points). After 3, 6 and 12 months of treatment, the dynamics of risk factors for progression was assessed: an increase in the severity of the risk factor meant +1, no change = 0, a decrease in the severity of the risk factor of -1.
Time Frame: Baseline and 3, 6 and 12 months
Population: ITT set
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
Scores
  Month 3 | -0.9 (0.9) | -0.7 (0.8)
  Month 6 | -0.7 (1.0) | -0.4 (0.8)
  Month 12 | -1.0 (1.0) | -0.6 (1.0)
Statistical Analysis 1: Comparison: Afalaza vs Placebo; Test type: Superiority; p = 0.0142, Mixed Models Analysis

10. Secondary Outcome: Number of Episodes of Acute Urinary Retention, Surgical Intervention During the Observation Period
Time Frame: 12 months
Population: ITT set
Measure: Number; unit: episodes
Arm/Group | Afalaza | Placebo
Number analyzed (Participants) | 119 | 117
episodes | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 12 months of therapy and 30 days after the end of the research
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=249, Safety Population)
Arm/Group | Afalaza | Placebo
Serious Adverse Events (participants affected / at risk) | 0/125 | 1/124
Other Adverse Events (participants affected / at risk) | 25/125 | 29/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afalaza (N=125) | Placebo (N=124)
Arthralgia/Meniscus injury/Meniscus operation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Resection of the medial meniscus and lateral meniscus. Resection of the mediapatulatory fold.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afalaza (N=125) | Placebo (N=124)
Prostatic specific antigen increased (Investigations) | 4 | 6
Epigastric pain (Gastrointestinal disorders) | 1 | 0
Right-sided inguinal hernia (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Chronic gastritis, exacerbation (Gastrointestinal disorders) | 0 | 1
Asthenia and Depressive weariness (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Labial herpes (Infections and infestations) | 1 | 0
Acute respiratory viral infection (Infections and infestations) | 9 | 10
Acute bronchitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 5
Vasomotor rhinitis chronic, exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Discomfort in the oropharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Сough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypertensive crisis, accompanied by headache and nausea (Vascular disorders) | 1 | 0
Chronic hemorrhoids, exacerbation (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes